CLINICAL TRIAL: NCT00815789
Title: Prevention of Cardiovascular Outcomes in African Americans With Diabetes
Brief Title: Cholesterol, Hypertension and Glucose Education Study
Acronym: CHANGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: The Kate B. Reynolds Charitable Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00006548; 64254 (Other Grant/Funding Number: Robert Wood Johnson Foundation); Pro00006548 (Other: Duke University IRB)
Record Dates: First submitted 2008-12-26; First posted 2008-12-30 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2014-07

CONDITIONS: Cardiovascular Disease; Diabetes
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): A nurse-administered intervention, which includes a behavioral and a medication management component. The intervention consists of very brief monthly telephone calls and occurs over 12 months. Upon request, participants may also be mailed additional supportive educational material to supplement phone intervention. They will also receive a letter clarifying medications reviewed with them during the nurse-administered intervention.
  Interventions: Behavioral: Tailored cardiovascular risk management (Nurse-administered )
- Control (No Intervention): Receive educational material about CVD reduction at baseline

INTERVENTIONS:
Behavioral: Tailored cardiovascular risk management (Nurse-administered ) — A nurse-administered intervention, which includes a behavioral and a medication management component. The intervention consists of very brief monthly telephone calls and occurs over 12 months. Upon request, participants may also be mailed additional supportive educational material to supplement phone intervention. They will also receive a letter clarifying medications reviewed with them during the nurse-administered intervention.
  Arms: Intervention

SUMMARY:
The goal of this study is to improve cardiovascular disease (CVD) and cholesterol in African Americans adults with diabetes by addressing the modifiable risk factors of systolic blood pressure (SBP), glycosylated hemoglobin (Hb A1c), and low-density lipoprotein cholesterol (LDL-C). We will evaluate the impact of a tailored CVD risk management intervention administered by nurses via the telephone. The intervention incorporates medication management and behavioral modification and will be tailored to the needs of vulnerable high risk subjects (e.g. African Americans, low socioeconomic status, low literate). It will be integrated into community clinics, thereby enhancing the potential for benefit and generalizability to other settings.

The primary hypothesis is that among African American subjects with diabetes, a nurse administered, tailored cardiovascular risk management intervention targeting both medication management and behavioral patient self-management will decrease SBP by 5 mmHg, Hb A1c by 0.5%, and LDL-C by 20 mg/dl over 12 months relative to the cardiovascular education-only control group.

DETAILED DESCRIPTION:
We will recruit eligible subjects who have an upcoming primary care visit with their primary care provider. Subjects will first be mailed letters, signed by a member of their own primary care team (in these clinics, patients are usually under the care of a team and not one physician) or the Clinic Medical Director in the absence of a primary team member, requesting their participation in the study. Subjects can call a toll-free number to request not to be contacted or if they have any questions (opt-out strategy similar to prior studies approved by Duke's IRB). The research assistant will contact the subject by telephone to explain the study, screen for eligibility, arrange an in-person meeting at the clinic to further describe the study, obtain informed consent and interview the subject. Enrollment will be scheduled at a time when individuals will already be coming to their clinic and all subsequent outcome assessment will be obtained from medical records (e.g., blood pressure, Hb A1c, and LDL-C, BMI) and secondary outcomes (e.g., behaviors will be obtained over the telephone).

Upon enrollment, each eligible, consenting subject will be surveyed about demographics, health behaviors (exercise, diet, medication compliance and treatment barriers), social and medical environment (experiences of discrimination, John Henryism, PHQ2, social support and stress, diabetes knowledge and communication). The entire interview would take approximately 60-90 minutes. If the interview cannot be completed at that time, we will ask permission to call the subject at home to complete the interview. After subjects have completed the measurement battery, they will be randomly assigned to be in one of the two groups. The entire study randomization will occur before patient enrollment begins and this will be maintained in a central site away from the enrollment site.

At either a 12-month follow-up visit or via a phone call, all subjects will once again be surveyed (30-60 minutes) to determine secondary outcome variables including changes in health behaviors, and adherence to recommended regimens. In addition, the cost-effectiveness of the intervention will be assessed at the conclusion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in one of the three primary care clinics for at least one year
* Diagnosis ICD (250.xx) in the prior year
* 18 years of age and older.

Exclusion Criteria:

* Hospitalized for a stroke, myocardial infarction, coronary artery revascularization in the past 6 months
* Receiving or planning to receive dialysis for end stage renal disease
* Diagnosis of metastatic cancer
* Active diagnosis of psychosis documented in medical record
* Does not have access to a telephone
* Refusal to provide informed consent
* Resident in nursing home or receiving home health care
* Severely impaired sight, hearing or speech
* Planning to leave the area prior to the anticipated end of participation
* Pregnant or planning to become or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2008-12; Primary Completion 2011-03 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in the outcome (SBP, Hb A1c, or LDL) from baseline to the 12 month evaluation. | 12 months

SECONDARY OUTCOMES:
Changes in CVD related health behaviors (e.g., aspirin use, medication adherence, exercise, and diet) as well as changes in stroke and CHD risk as assessed by the UPKDS risk engine | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hayden B Bosworth, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Health Care System, Durham, North Carolina, United States

REFERENCES:
- [Derived] Crowley MJ, Powers BJ, Olsen MK, Grubber JM, Koropchak C, Rose CM, Gentry P, Bowlby L, Trujillo G, Maciejewski ML, Bosworth HB. The Cholesterol, Hypertension, And Glucose Education (CHANGE) study: results from a randomized controlled trial in African Americans with diabetes. Am Heart J. 2013 Jul;166(1):179-86. doi: 10.1016/j.ahj.2013.04.004. Epub 2013 May 17. PMID 23816038